CLINICAL TRIAL: NCT00482560
Title: Analgesic Effect of Breast Feeding vs Sucrose in Neonatal Screening
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Agnelli Hospital, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRN19341
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2007-06-29 (Estimated); Status verified 2007-06

CONDITIONS: Pain
Keywords: Sucrose; Breastfeeding; Heel lance
MeSH Terms: conditions — Pain; Breast Feeding | interventions — Lactation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sucrose solution 30%1 ml
Behavioral: Breastfeeding

SUMMARY:
The purpose of this study is to compare the antinociceptive effect of 1 ml of 30% sucrose solution vs breastfeeding on neonatal screening heel lance

DETAILED DESCRIPTION:
Blood sampling heel lance for neonatal screening is the most frequent painful manoeuvre in Neonatal Units in healthy neonates.

Some techniques showed efficacy evidence in reducing pain response: sucrose solutions, breastfeeding during blood sampling, topical local anaesthetics.

A Cochrane Review in 2004 recommends the administration of sucrose 0.24-0.48 g (1-2 ml of 24% sucrose solution). It reduces PIPP scale rate about 20%.

Our purpose is to compare the antinociceptive effect of 1 ml 30% sucrose solution administered 2 minutes before heel lancing vs blood sampling heel lance during breastfeeding.

PIPP scale is a validated 7-indicator scale for the assessment of procedural pain in preterm and term neonates.

Informant consent was asked parents during consultation by a Pediatrician of the Neonatal Unit of the Hospital in the last months of pregnancy.

After parent written consent was obtained, 100 three day old neonates were randomized for treatment A (breastfeeding) or B (sucrose solution administration). The nurse opened consecutively numbered envelopes.

Timing of operators: Group A Breastfeeding

* The heel of neonate was warmed up by a glove full of water at 40° C for 2 minutes.
* Monitoring of Oxygen Saturation and Heart Rate.
* The neonate was breastfed by the mother till the nurse watched a continuous active suction.
* Administration of first phase of PIPP scale (15 seconds before heel lance).
* Digital Voice Record started
* Heel Lance with an automated piercing device .
* Squeezing for blood sampling till filling 4 catch basins for neonatal screening. If necessary a new heel lance was practiced.
* Administration of the second phase of PIPP scale.
* Record of duration of blood sampling and collateral effects
* Stop Digital Voice Recording

Group B Sucrose administration

* The neonate was laid on a baby-changing table.
* The heel of neonate was warmed up by a gloves full of water a 40° C for 2 minutes.
* Oral administration of 1 ml of 30% sucrose solution.
* Monitoring of Oxygen Saturation and Heart Rate.
* Administration of first phase of PIPP scale (15 seconds before heel lance).
* Digital Voice Record starts
* Heel Lance with an automated piercing device.
* Squeezing for blood sampling till filling 4 catch basins for neonatal screening. If necessary a new heel lance was practiced.
* Administration of the second phase of PIPP scale.Record of duration of blood sampling and collateral effects.
* Stop Digital Voice Recording

Blood sampling was practiced by skilled pediatric nurses. Registration of data, PIPP scale, voice record was made by a second operator, blind to the pur pose of the study.

A third blind operator collected paper data and checked voice record (outcome cry behaviour).

ELIGIBILITY:
Inclusion Criteria:

* Term neonates, gestational age 37-42 weeks
* Apgar >= 7
* Not fed in the last 30 minutes
* Informant consent

Exclusion Criteria:

* Congenital malformation
* Born in Caesarian Section in General Anaesthesia
* Maternal use of opioids
* Administration of Naloxone, Phenobarbital in the previous 48 hours
* Impossibility of breastfeeding

Ages: 2 Days to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2007-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Premature Infant Pain Profile (PIPP) scale rate (0-21) | 15 seconds before and Within 30 seconds after heel lance

SECONDARY OUTCOMES:
Heart Rate Increase | within 30 seconds after heel lance
Oxygen Saturation decrease | within 30 seconds after heel lance
Duration of first cry | within 2 minutes after heel lance
Percentage of crying time | within 2 minutes after heel lance
Percentage of crying time | During blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Codipietro, MD, Principal Investigator — University of Turin Department of Paediatric Science Doctorate in Experimental Pediatry; Alberto Ponzone, MD, Study Chair — University of Turin Department of Paediatric Science Doctorate in Experimental Pediatry
Locations (1):
- Agnelli Hospital ASL 10, Pinerolo, Torino, Italy

REFERENCES:
- [Background] Stevens B, Yamada J, Ohlsson A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2004;(3):CD001069. doi: 10.1002/14651858.CD001069.pub2. PMID 15266438
- [Background] Carbajal R, Veerapen S, Couderc S, Jugie M, Ville Y. Analgesic effect of breast feeding in term neonates: randomised controlled trial. BMJ. 2003 Jan 4;326(7379):13. doi: 10.1136/bmj.326.7379.13. PMID 12511452
- [Background] Shah PS, Aliwalas LI, Shah V. Breastfeeding or breast milk for procedural pain in neonates. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD004950. doi: 10.1002/14651858.CD004950.pub2. PMID 16856069
- [Background] Ballantyne M, Stevens B, McAllister M, Dionne K, Jack A. Validation of the premature infant pain profile in the clinical setting. Clin J Pain. 1999 Dec;15(4):297-303. doi: 10.1097/00002508-199912000-00006. PMID 10617258
- [Derived] Codipietro L, Ceccarelli M, Ponzone A. Breastfeeding or oral sucrose solution in term neonates receiving heel lance: a randomized, controlled trial. Pediatrics. 2008 Sep;122(3):e716-21. doi: 10.1542/peds.2008-0221. PMID 18762508